CLINICAL TRIAL: NCT03299816
Title: Community-Based Dietary Approach for Hypertensive African Americans With Chronic Kidney Disease
Brief Title: Five, Plus Nuts and Beans for Kidneys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00122943; 1U01MD010550-01 (NIH)
Record Dates: First submitted 2017-09-18; First posted 2017-10-03 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Chronic Kidney Disease; Hypertension; Albuminuria; African Americans
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Albuminuria

STUDY DESIGN:
Intervention Model Description: Single center, randomized controlled trial with two parallel arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Shopping DASH group (S-DASH) (Active Comparator): The Self-Shopping DASH group will receive printed patient-centered materials on the DASH diet and chronic kidney disease. Participants will also receive $30/week allowance for the purchase of food and drinks of their choosing from a local grocer (Klein's ShopRite stores of Maryland) during the first four months. During the remainder of the study (months 5-12), the participants in this group will be asked to continue to follow the dietary advice provided but will not receive the food allowance.
  Interventions: Behavioral: Self-Shopping DASH group (S-DASH)
- Coaching DASH group (C-DASH) (Experimental): The C-DASH group intervention will be a patient-tailored program, delivered by a study coach that is trained by a dietitian, which emphasizes key self-management behaviors - diet and self-monitoring. This group will receive advice from the study coach and purchase $30 worth of fresh fruits, vegetables, nuts and beans that are high in potassium on a weekly basis for the first four months.
  Interventions: Behavioral: Coaching DASH group (C-DASH)

INTERVENTIONS:
Behavioral: Coaching DASH group (C-DASH) — Participants assigned to the C-DASH diet advice group will be provided $30/week worth of fruits, vegetables, nuts and beans ordered through the study coach and delivered to a community location to reach a certain goal of potassium intake (months 0-4). During phase 2 of the study (months 5-12), a study coach will continue telephonic contact with the participants to set goals for following a DASH-like diet without the weekly food allowance.
  Other Names: Coaching DASH diet advice group (C-DASH)
  Arms: Coaching DASH group (C-DASH)
Behavioral: Self-Shopping DASH group (S-DASH) — Participants will be given a brochure containing information about the DASH diet which will be reviewed with a study team member. In months 1-4, participants will receive a gift card equivalent to a weekly allowance of $30 to Klein's ShopRite stores of Maryland for purchases of food and beverages of their choice. During phase two (months 5-12), they will be asked to continue following a DASH-like diet but will not receive a gift card for purchases.
  Other Names: Self-Shopping DASH diet advice Group (S-DASH)
  Arms: Self-Shopping DASH group (S-DASH)

SUMMARY:
This Five, Plus Nuts and Beans for Kidneys Study is a single center, randomized controlled trial with 2 parallel arms testing the hypothesis that delivery of nutritional advice to adopt a Dietary Approaches to Stop Hypertension (DASH)-like diet and $30/week worth of fruits, vegetables, nuts and beans tailored to personal choices and availability in neighborhood stores, will reduce kidney damage in African Americans with hypertension and chronic kidney disease.

DETAILED DESCRIPTION:
This study will test the effectiveness of dietary advice delivered by a study coach and assistance with weekly online ordering of $30/week worth of potassium rich foods delivered by a local grocer to a community location for reducing urinary albumin excretion among African Americans with hypertension and chronic kidney disease. Participants will be recruited from primary care clinics in Baltimore, MD.

150 African American adults diagnosed with hypertension and with mild/moderate chronic kidney disease based on the presence of albuminuria will be randomly assigned to one of two arms for 12 months. There are 2 phases of the study. In Phase 1 (months 1-4), one study arm will consist of minimal guidance from the study team and a weekly allowance of $30 dollars to purchase food and drinks of their choosing from a local grocer. During Phase 1, the second arm of the study will receive dietary guidance from the study coach and assistance with ordering and purchasing $30/week worth of high potassium foods from the same local grocer. In Phase 2 (months 5-12) neither study arm will receive a food allowance, however the second arm will receive telephonic visits and dietary advice from the study coach.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African American race
* Age 21 years or older
* Clinical diagnosis of hypertension and have a urine Albumin-Creatinine Ratio (ACR) of ≥30 mg/g with or without estimated Glomerular Filtration Rate (GFR) 30-59 ml/min/1.73m2.
* Must be under regular care with their Johns Hopkins Community Physicians (JHCP) or Johns Hopkins Outpatient Center (JHOC) physician (seen within the past 12 months).
* Must have a systolic blood pressure of <=160 mmHg and a diastolic blood pressure of <=100 mmHg (average of two visits)
* Be on stable doses of antihypertensive medications for a minimum of two months prior to randomization.

Exclusion Criteria:

* Cardiovascular (CV) event within 6 months
* Chronic disease that might interfere with trial participation (e.g. stage 4 or 5 Chronic Kidney Disease, Estimated Glomerular Filtration Rate <30 ml/min/1.73m2)
* Unwillingness or inability to adopt a DASH-like diet
* Consumes over 14 alcoholic drinks per week
* Poorly controlled diabetes (Hemoglobin A1c >9%).
* Patients with a serum potassium >4.6 milliequivalent (mEq) /L45
* Urine ACR ≥ 1,000 mg/g

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deidra Crews, MD, ScM, Principal Investigator — Johns Hopkins University
Locations (1):
- East Baltimore Medical Campus, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share the Statistical Analysis Plan and Study Protocol.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after one year after final data collection.
Access Criteria: Will release de-identified information per request via Johns Hopkins agreement.

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: 4-month Intervention Period
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Started | 70 | 72
Completed | 69 | 72
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Phase 2: 12-month Follow-up Period
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Started | 52 (The number of eligible C-DASH participants included 53 who were randomized prior to 2021, minus 1 who dropped out during Phase 1. Seventeen C-DASH participants who were randomized in 2021 were invited to participate in Phase 1 only and were not included in Phase 2 of this study.) | 56 (The number of eligible S-DASH participants included 56 who were randomized prior to 2021. Sixteen S-DASH participants who were randomized in 2021 were invited to participate in Phase 1 only and were not included in Phase 2 of this study.)
Completed | 49 | 53
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH) | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (13.7) | 62.7 (11.7) | 61.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 40 | 90
  Male | 20 | 32 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 69 | 71 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 69 | 71 | 140
  White | 0 | 0 | 0
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 72 | 142
Baseline Urinary albumin-to-creatine (ACR) [Mean (Inter-Quartile Range); unit: mg/g] | 99.8 [49.0 to 234.5] | 98.8 [47.3 to 236.5] | 99.5 [4.08 to 234.5]
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.1 (14.4) | 130.8 (12.8) | 129.4 (13.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72.3 (10.6) | 74.4 (11.2) | 73.3 (10.9)
Diabetes (Self-report) [Count of Participants; unit: Participants] | 32 | 31 | 63
Urinary albumin-to-creatine ratio category [Count of Participants; unit: Participants]
  <30 mg/g | 6 | 6 | 12
  30 to <300 mg/g | 53 | 51 | 104
  >=300 mg/g | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Albumin Excretion From Baseline to 4 Months
Description: Urine samples will be collected for ACR (albumin-to-creatinine ratio).
Time Frame: Baseline, 4 months
Population: For C-DASH, 3 participants were excluded from analysis: 1 withdrew from the study and 2 were lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 67 | 72
mg/g | -28.6 (12.0) | -5.6 (11.6)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.17, Mixed effects regression — The a priori threshold for statistical significance was <0.05; Urinary albumin-to-creatinine ratio (ACR) was not normally distributed and was natural log transformed for analyses

2. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to 4 Months
Description: Daytime systolic blood pressure monitoring will be determined using OMRON 907-xl
Time Frame: Baseline,4 months
Population: For C-DASH, 4 participants were excluded from analysis: 1 withdrew from the study, 2 were lost to follow-up, and 1 was due to measurement error. For S-DASH, 5 participants were excluded: 4 were due to measurement error, and 1 due to an out-of-range baseline reading.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 66 | 67
mm Hg | -1.4 (1.8) | 0.9 (1.7)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.36, Mixed effects regression — The a priori threshold for statistical significance was <0.05

3. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to 12 Months
Description: Daytime systolic blood pressure monitoring will be determined using OMRON 907-xl
Time Frame: Baseline, end of study (approximately 12 months)
Population: For C-DASH, 9 participants were excluded from analysis: 1 withdrew from Phase 2 of the study, 3 were lost to follow-up, 1 due to measurement error, 1 moved out of state, and 3 were restricted from providing in-person data collection due to the COVID-19 pandemic. For S-DASH, 12 participants were excluded: 4 were lost to follow-up, 5 due to measurement error, and 3 were restricted from in-person data collection due to the pandemic.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 43 | 44
mm Hg | 1.5 (2.3) | -1.6 (2.3)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.33, Mixed effects regression — The a priori threshold for statistical significance was <0.05

4. Secondary Outcome: Change in Urinary Albumin Excretion From Baseline to 12 Months
Description: Urine samples will be collected for ACR (albumin-to-creatinine ratio).
Time Frame: Baseline, end of study (approximately 12 months)
Population: For C-DASH, 7 participants were excluded from analysis: 1 withdrew during Phase 2 of the study, 2 were lost to follow-up, and 4 were restricted from providing in-person data collection due to the COVID-19 pandemic. For S-DASH, 8 participants were excluded: 3 were lost to follow-up, 1 sample was lost due to lab error, and 4 were restricted due to the pandemic.
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 45 | 48
mg/g | -11.5 (14.1) | -1.4 (13.7)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.61, Mixed effects regression — The a priori threshold for statistical significance was <0.05; Urinary albumin-to-creatinine ratio (ACR) was not normally distributed and was natural log transformed for analyses

5. Other Pre Specified Outcome: Change in Urinary Albumin Excretion From Baseline to 1 Month
Description: Urine samples will be collected for ACR (albumin-to-creatinine ratio).
Time Frame: Baseline, 1 month
Population: For C-DASH, 3 participants were excluded from analysis: 1 withdrew from the study, and 2 were lost to follow-up. For S-DASH, 1 participant was excluded from analysis due to an invalid urine sample.
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 67 | 71
mg/g | -14.8 (10.1) | -19.6 (9.8)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.73, Mixed effects regression — The a priori threshold for statistical significance was <0.05; Urinary albumin-to-creatinine ratio (ACR) was not normally distributed and was natural log transformed for analyses

6. Other Pre Specified Outcome: Change in Systolic Blood Pressure From Baseline to 1 Month
Description: Daytime systolic blood pressure monitoring will be determined using OMRON 907-xl
Time Frame: Baseline, 1 month
Population: For C-DASH, 7 participants were excluded from analysis: 1 withdrew from the study, 2 were lost to follow-up, and 4 were due to measurement error. For S-DASH, 4 participants were excluded: 3 were due to measurement error, and 1 due to an out-of-range at baseline reading.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
Number analyzed (Participants) | 63 | 68
mm Hg | -1.1 (1.6) | -0.3 (1.5)
Statistical Analysis 1: Comparison: Coaching DASH Group (C-DASH) vs Self-Shopping DASH Group (S-DASH); Test type: Superiority; p = 0.75, Mixed effects regression — The a priori threshold for statistical significance was <0.05

ADVERSE EVENTS:
Time Frame: The first 108 randomized participants: 1 year; The remaining 33 randomized participants: 4 months
Arm/Group | Coaching DASH Group (C-DASH) | Self-Shopping DASH Group (S-DASH)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/72
Serious Adverse Events (participants affected / at risk) | 7/70 | 7/72
Other Adverse Events (participants affected / at risk) | 10/70 | 16/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coaching DASH Group (C-DASH) (N=70) | Self-Shopping DASH Group (S-DASH) (N=72)
Abdominal Pain (Gastrointestinal disorders) | 1 (4) | 0 (0)
Cardiac Catheterization (Surgical and medical procedures) | 0 (0) | 1 (1)
Angioneurotic edema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — due to lisinopril
Acute kidney failure (Renal and urinary disorders) | 1 (1) | 0 (0) — possibly due to Lisinopril
Cerebral infarction, unspecified (Vascular disorders) | 0 (0) | 1 (1)
Chronic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus with ketoacidosis (Endocrine disorders) | 1 (1) | 0 (0)
Mechanical complication of ventricular intracranial (communicating) shunt (Nervous system disorders) | 1 (1) | 0 (0)
Moderate persistent asthma with (acute) exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Angina pectoris (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm and dissection (Vascular disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain, unspecified (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-ST elevation myocardial infarction (Vascular disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thrombophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Type 2 Subsequent non-ST elevation myocardial infarction (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coaching DASH Group (C-DASH) (N=70) | Self-Shopping DASH Group (S-DASH) (N=72)
Hypertensive Urgency (Vascular disorders) | 3 (4) | 10 (14) — BP >= 160/100
Hypokalemia (Metabolism and nutrition disorders) | 7 (9) | 6 (6)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic restricted in-person research activities for ~6 months, which impacted trial conduct in two ways: (1) 8 of the participants randomized at the onset of the pandemic did not return when restrictions on in person research were lifted. They were excluded from the final sample size. (2) Upon resuming in-person activities, the protocol was modified to Phase 1 only for the 33 participants who were randomized in 2021, so that the trial could be completed within the funding period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03299816/Prot_SAP_004.pdf